CLINICAL TRIAL: NCT04039256
Title: Efficacy And Safty of Heartech® Left Ventricular Partitioning Device In Treating Heart Failure Post Myocardial Infarction (Phase II Clinical Trial: The Partical Study)
Brief Title: Phase II Clinical Trial of Percutaneous Ventricular Restoration Using Heartech® Device Preventing Heart Failure Post Myocardial Infarction (The Partical Study)
Acronym: Partical
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhang Qi, MD, Chief of Cardiology Department, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-20190728
Record Dates: First submitted 2019-07-28; First posted 2019-07-31 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Efficacy, Safty, Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PVR implantation group (Experimental): Patients enrolled receive PVR intervention
  Interventions: Device: percutaneous ventricular restoration using heartech® device

INTERVENTIONS:
Device: percutaneous ventricular restoration using heartech® device — Patients who are confirmed suitability by imaging analysis, receive heartech® left ventricular partitioning device implantation.

SUMMARY:
This is a prospective, multi-center, single-group, target-value clinical study. The primary safety end points are major adverse cardiovascular events (MACCE) 30 days after device implantation.

The primary efficacy end point is the end of left ventricular systolic volume index (LVESVI) reduction at 6 month.

The secondary observational end points includes immediate success rate of the procedure, all-cause mortality, cardiac death, rehospitalization rates and MACCE occurrence rate within 12 month. Besides, left ventricular end systolic volume index (LVESVI) change at 30 days,12 months, left ventricular ejection fraction (LVEF), left ventricular end-diastolic volume index (LVEDVI), 6 minutes walk test, heart function evaluation (NYHA classification) and quality of life (EQ-5D) at 30 days, 6 months, 12 months will also be evaluated.

After statistical hypothesis and sample size estimation, the sample size of this clinical trial was 117 cases. All subjects were followed up 30 days, 6 months and 12 months after implantation of the Heartech® left ventricular partitioning device. All relevant clinical data were managed by professional data management center, and all relevant clinical data were statistically analyzed by third-party statistical center.

DETAILED DESCRIPTION:
MACCE includes all-cause death, myocardial infarction, stroke and any elective or emergency cardiac or thoracic aortic surgery or catheter-based interventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* BMI<40;
* left ventricular ejection fraction ≤45% and ≥20%;
* patients with left ventricular end-systolic volume index (ESVI) ≥50mL/m2;
* transthoracic ultrasound showed contradictory motion of the left ventricle after myocardial infarction;
* 60 days prior to anterior wall myocardial infarction with ischemic heart failure (NYHA grade II to "not hospitalized" grade IV);
* the left ventricle must have the appropriate anatomic structure (size and shape) which is confirmed by cardiac CT and left ventricular angiography to implant the appropriate Heartech® device;
* agree to receive reasonable treatment according to current ACC/AHA and Chinese guidelines for heart failure diagnosis and treatment;
* the subjects or their legal representatives are informed of the nature of this study and agree to participate in all the terms of this study, sign the informed consent approved by the ethics committee, agree to accept the postoperative treatment plan and follow-up requirements, and can complete the examination of follow-up.

Exclusion Criteria:

* patients whose left ventricular anatomy is not suitable for Heartech® occlusal device implantation;
* the abnormal ventricular wall movement not contains the anterior wall of the left ventricle, the apex of the left ventricle and the ventricular septum;
* patients with thrombosis in the left ventricle;
* mitral stenosis or regurgitation (tricuspid, aortic or mitral) > 2+ (moderate);
* recent (within 6 month) cerebrovascular accident (CVA) or transient ischemic attack (TIA);
* end-stage renal disease requiring long-term dialysis, episodic sepsis or active phase endocarditis;
* life expectancy at admission < 1 year;
* known allergy to aspirin, heparin, warfarin, Nitinol (alloys of titanium and nickel) or contraindications, or sensitivity to contrast agents;
* cardiogenic shock occurred within 72 hours before procedure;
* pregnancy or planned pregnancy during the study period;
* participated in clinical trials of other drugs or medical devices during the same period;
* the researcher judged that the patient had poor compliance and could not complete the study as required;
* other conditions considered unsuitable for participation in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACCE [primary safety] | 30 days
  major adverse cardiovascular events (MACCE)
LVESVi Reduction [primary efficacy] | 6 month
  left ventricular systolic volume index (LVESVi) reduction

SECONDARY OUTCOMES:
Procedure Success | immediate
  success rate of the procedure
Mortality | 12 month
  all-cause mortality rate
Cardiac death | 12 month
  cardiac death rate
Rehospitalization | 12 month
  rehospitalization rate
Incidence of MACCE | 12 month
  MACCE occurrence rate
LVESVi Reduction | 12 month
  left ventricular end systolic volume index (LVESVi) change
LVEDVi Reduction | 12 month
  left ventricular end-diastolic volume index (LVEDVi)
LVEF change | 12 month
  left ventricular ejection fraction (LVEF) detected by echocardiography
Cardiac function | 12 month
  cardiac function evaluation (NYHA classification)
Walk tolerance | 12 month
  6 minutes walk test
life quality | 12 month
  quality of life (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Fenghua Ding, MD. Ph.D., Study Director — Cardiovascular research instittion, Shanghai Jiao Tong University
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu Z, Yu J, Xu K, Tang Y, Fang Y, Gu J, Gu S, Ding F, Modine T, Zhang R. First-in-man study of Heartech(R) percutaneous left ventricular partitioning device for treatment of heart failure postmyocardial infarction. Catheter Cardiovasc Interv. 2019 Nov 15;94(6):845-853. doi: 10.1002/ccd.28366. Epub 2019 Jun 23. PMID 31231944